CLINICAL TRIAL: NCT03961269
Title: Frequency and Presentations of Chronic Pain Following Breast Cancer Surgery: An Observational Study in a Tertiary Care Hospital of Pakistan
Status: Completed | Type: Observational
Sponsor: Ali Sarfraz Siddiqui (Other)
Responsible Party: Sponsor-Investigator, Ali Sarfraz Siddiqui, Assistant Professor, Aga Khan University
Organization: Aga Khan University (Other)
Other Study IDs: 4257-Ane-ERC-16
Record Dates: First submitted 2019-05-16; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer Female; Chronic Pain
Keywords: Breast cancer surgery; Persistent pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to evaluate the frequency and presentations of chronic persistent pain in patients after breast cancer surgery at our tertiary care hospital. Results of this study will help us to understand the magnitude of problem in our population and making institutional guidelines for appropriate management of such patients.

DETAILED DESCRIPTION:
After approval from the Departmental Research Committee and Institutional Ethical Review Committee all adult female patients with known carcinoma of breast who are scheduled for elective definitive breast cancer surgery (Mastectomy) from 1st July 2016 to 30th December 2016 will be enrolled in this audit. Inclusion of patients will be done once operative procedure is finalized and consent taken in breast clinic. Those patients who did not give consent and those patients who need reoperation on same side for recurrence of cancer or any reason will be excluded from this study.

Data will be obtained from patient's medical record, interview of patient on follow up visit at breast clinic and telephonic communication with patient. Variables have been defined and a special form has been designed for data collection. All patients will be followed for next three months and those who have persistent pain will be followed for six months after operation.

Follow up information will be obtained from patient visiting breast clinic. For any missing data patient's medical records will be reviewed and patient will be contacted to know if they have chronic post-surgical pain or not. Audit forms will be filled by authors according to their availability. The primary investigator or author at breast clinic will keep all forms for safe record keeping which shall later be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* all adult female patients with known carcinoma of breast who are scheduled for elective definitive breast cancer surgery (Mastectomy)

Exclusion Criteria:

* Those patients who did not give consent and those patients who need reoperation on same side for recurrence of cancer or any reason will be excluded from this study.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All female patient with breast cancer
Study Population: all adult female patients with known carcinoma of breast who are scheduled for elective definitive breast cancer surgery (Mastectomy)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
To determine the frequency of persistent pain in patients after breast cancer surgery | 3 to 6 months
  After breast cancer surgery, patients were followed for next 3 months and those patients who developed persistent pain were followed for up to 6 months via pre designed questionnaire

SECONDARY OUTCOMES:
To observe the distribution and characteristics of pain in these patients. | 3 to 6 months
  After breast cancer surgery, patients were followed to observe the distribution and characteristics of pain on pre-designed questionnaire

IPD SHARING:
Plan to Share IPD: No